CLINICAL TRIAL: NCT02243943
Title: Effect of Neuromuscular Blockade Reversal With Sugammadex on Oxygenation, Pain and Arousal States in the Post Anesthesia Care Unit
Brief Title: Effect of Neuromuscular Reversal With Sugammadex on Postoperative Recovery Profile
Acronym: Neuropa
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Albert Dahan, Prof. Dr. A. Dahan, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL34186.058.10; NL34186.058.10 (Other: LUMC)
Record Dates: First submitted 2014-09-12; First posted 2014-09-18 (Estimated); Results first posted 2016-08-25 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2016-12

CONDITIONS: Postoperative Respiratory Condition
Keywords: Neuromuscular block; neuromuscular reversal; postoperative conditions; respiratory failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugammadex (Experimental): Subjects in this arm will be reversed with sugammadex 2-4 mg/kg
  Interventions: Drug: Sugammadex
- neostigmine (Active Comparator): subjects in this arm will be reversed with neostigmine 1.0-2.5 mg and atropine 0.5-1.0mg
  Interventions: Drug: Neostigmine

INTERVENTIONS:
Drug: Sugammadex
  Other Names: Bridion
  Arms: Sugammadex
Drug: Neostigmine
  Other Names: Prostigmin
  Arms: neostigmine

SUMMARY:
Suboptimal reversal of neuromuscular blockage after surgery is possibly related to unfavorable postoperative respiratory conditions and elevated pain levels. Rapid and complete reversal of neuromuscular block was not possible untill sugammadex was discovered. The investigators hyposthesise that reversal with sugammadex leads to favorable postoperative respiratory conditions and less pain compared to reversal with neostigmine.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years
* - BMI < 35
* -ASA class I- III
* -Patients scheduled for surgery requiring general anesthesia with the use of NMBA's

  * Patients with ability to give oral and written informed consent

Exclusion Criteria:

* Failure to meet the inclusion criteria

  * -Known or suspected neuromuscular disorders impairing neuromuscular function
  * -Allergies to muscle relaxants, anesthetics or narcotics
* A (family) history of malignant hyperthermia

  * -Women who are or may be pregnant or are currently breast feeding
  * -Contraindications for the use of neostigmine
* Intestinal obstruction,
* COPD GOLD 4

  * -Abnormal heart rhythm (eg. bradycardia: < 40/min);
  * -Surgery requiring neuraxial anesthesia / analgesia
  * -Preoperative cognitive dysfunction or mental disabilities
  * -Preexistent significant pulmonary disease with preoperative SpO2 < 90%
  * -Preoperative ICU treatment / intubation (ICU patient);
  * -Need for postoperative ICU treatment or ventilation;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Dahan, MD, PhD, Professor, Principal Investigator — Leiden Medical University
Locations (1):
- Leiden Medical University, Leiden, South Holland, Netherlands

RESULTS

PARTICIPANT FLOW:
Groups:
- Sugammadex: Subjects in this arm will be reversed with sugammadex 2-4 mg/kg
  Sugammadex
- Neostigmine: subjects in this arm will be reversed with neostigmine 1.0-2.5 mg and atropine 0.5-1.0mg
  Neostigmine
Period: Overall Study
Arm/Group | Sugammadex | Neostigmine
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugammadex | Neostigmine | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Median (Full Range); unit: years of age] | 55 [27 to 72] | 55 [19 to 94] | 55 [19 to 94]
Gender [Count of Participants; unit: Participants]
  Female | 27 | 24 | 51
  Male | 23 | 26 | 49

OUTCOME MEASURES:

1. Primary Outcome: Mean Lowest Saturation
Description: Mean saturation is the mean value of the beat-to-beat Hb-oxygen saturation measured by finger pulse oximeter as measured in the first 45 min in the recovery room following surgery
Time Frame: 45 minutes post surgery
Measure: Mean (95% Confidence Interval); unit: percentage of oxygen saturation
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 50 | 50
percentage of oxygen saturation | 96.8 [96.1 to 97.4] | 93.3 [91.9 to 94.7]

2. Secondary Outcome: Pain
Description: using the 1-10 numeric rating scale
Time Frame: 45 minutes post surgery
Measure: Mean (95% Confidence Interval); unit: Numeric rating scale. 1(low)-10(maximum)
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 50 | 50
Numeric rating scale. 1(low)-10(maximum) | 3.0 [2.3 to 3.7] | 3.2 [2.4 to 4.0]

3. Secondary Outcome: Sedation
Description: using the Leiden observer alertness score (1 alert - 5 sedated)
Time Frame: 45 minutes post surgery
Measure: Mean (95% Confidence Interval); unit: sedation scale (1 alert - 5 sedated)
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 50 | 50
sedation scale (1 alert - 5 sedated) | 1.4 [1.2 to 1.6] | 1.4 [1.2 to 1.6]

ADVERSE EVENTS:
Arm/Group | Sugammadex | Neostigmine
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes